CLINICAL TRIAL: NCT01781390
Title: A Prospective, Double-Blind, Randomized, Placebo-controlled Clinical Trial of Intracoronary Infusion of Mesenchymal Precursor Cells (MPC) in the Treatment of Patients With ST-Elevation Myocardial Infarction
Brief Title: Safety Study of Allogeneic Mesenchymal Precursor Cell Infusion in Myocardial Infarction
Acronym: AMICI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mesoblast, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mesoblast, Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANG.AMI-IC001; 2010-020497-41 (EudraCT Number)
Record Dates: First submitted 2013-01-14; First posted 2013-02-01 (Estimated); Results first posted 2022-01-18 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute Myocardial Infarction; STEMI; Heart Attack; AMI; Stem Cells
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Placebo (Placebo Comparator): Participants received matching-placebo solution 2 milliliters per minute (mL/min) infused Intracoronary for 60 min including line flush [0 Mesenchymal Precursor Cells (MPCs)/min] on Day 0.
  Interventions: Other: Placebo
- Mesenchymal Precursor Cells (MPC) 12.5 M (Experimental): Participants received MPC 12.5 solution 2 mL/min infused Intracoronary for 60 min including line flush (2.5x10^5 MPCs/min) on Day 0.
  Interventions: Biological: Mesenchymal Precursor Cells (MPC) 12.5 M
- Mesenchymal Precursor Cells (MPC) 25 M (Experimental): Participants received MPC 12.5 solution 2 mL/min infused Intracoronary for 60 min including line flush (5.0x10^5 MPCs/min) on Day 0.
  Interventions: Biological: Mesenchymal Precursor Cells (MPC) 25 M

INTERVENTIONS:
Other: Placebo — Matching placebo solution for infusion.
  Arms: Placebo
Biological: Mesenchymal Precursor Cells (MPC) 12.5 M — MPC 12.5 M solution for infusion.
  Arms: Mesenchymal Precursor Cells (MPC) 12.5 M
Biological: Mesenchymal Precursor Cells (MPC) 25 M — MPC 25 M solution for infusion.
  Arms: Mesenchymal Precursor Cells (MPC) 25 M

SUMMARY:
This was a double-blind, randomized, placebo-controlled study that was designed to enroll a total of 225 participants with de novo anterior wall acute ST-segment elevation myocardial infarction (STEMI) due to a lesion of the left anterior descending coronary artery undergoing percutaneous coronary intervention (PCI). Eligible participants were to be enrolled and undergo revascularization of the culprit left anterior descending (LAD) coronary artery. The interventional procedure included as dose ranging assessment of intracoronary (IC) delivery of MPC or placebo infused into the stented coronary artery. This study compared two doses of MPCs and a placebo control group. Study participants were randomly assigned in 1:1:1 fashion to receive either 12.5 Million or 25 Million MPCs or placebo (saline). Initially, each group was designed to have approximately 75 patients per treatment group. The Primary Objective of the study was to determine the safety and feasibility of IC infusion of investigational MPCs in this acute STEMI population.

The Primary Objective of the study was to determine the safety and feasibility of IC infusion of investigational MPCs in this acute STEMI population. Feasibility of the infusion of the investigational agent was assessed by measurement of thrombolysis in myocardial infarction (TIMI) flow and perfusion (1) immediately prior to, (2) during (after approximately 50% of total investigational agent volume infused) and (3) following the investigational agent infusion after successful PCI and stenting. There was no evidence of clinically important coronary microvascular obstruction related to infusion of the investigational agent.

DETAILED DESCRIPTION:
This was a prospective, double-blind, randomized, placebo-controlled study that was designed to enroll approximately 225 participants with de novo anterior STEMI due to a lesion involving the proximal-mid LAD coronary artery who undergo primary PCI at approximately 45 clinical study sites. However, due to difficulty in consenting participants and operationalizing the protocol under the emergency environment of an acute STEMI, it became clear that a major protocol amendment would be required. Accordingly, the protocol was adjusted to randomize 105 participants (35 per treatment group) at 25 clinical study sites. This 53% reduction in participants from the original protocol allowed preliminary evaluations of safety and feasibility.

Potential participants who were in the midst of experiencing an acute anterior wall STEMI, where increased time to coronary revascularization is known to correlate with the extent of subsequent myocardial necrosis, were approached by a study site investigator prior to PCI to determine the participant's interest to participate in a stem cell investigational trial. This required the patient to sign an informed consent permitting both the PCI procedure and participation in the trial. Participants who agreed to participate in the AMICI study and had a successful and uneventful PCI and stenting of the culprit LAD lesion performed were then randomized to one of the three treatment groups. The randomization and treatment assignment were obtained using an interactive voice-response system (IVRS/interactive web response system [IWRS]). The following stratification for duration of cardiac ischemia was performed to ensure balanced randomization across the treatment groups:

* ≤2 hours
* >2 hours to ≤6 hours
* >6 to ≤12 hours

Eligible participants received intracoronary delivery of the assigned treatment infused via a microcatheter into the stented culprit artery.

After approximately 50% of the intracoronary infusion of investigational treatment was completed, an angiographic determination of coronary flow was performed. The following guidelines were used to determine if the remaining investigational agent should be infused:

The study infusion should have been continued if TIMI 2 or TIMI 3 flow was present in the absence of ALL of the following;

* Sustained hypotension not responsive to fluid administration;
* Clinical signs/symptoms indicating an acute cerebrovascular event;
* Re-elevation of ST-segments if previously resolved with PCI;
* Onset of the participant's symptoms of myocardial ischemia unresponsive to appropriate interventions;
* Two episodes of sustained ventricular tachycardia (VT)/ventricular fibrillation (VF) requiring cardioversion (infusion can continue if a single episode of sustained VT/VF requiring cardioversion occurred).

Feasibility of the infusion of the investigational agent was assessed by measurement of TIMI flow and perfusion (1) immediately prior to, (2) during (after approximately 50% of total investigational agent volume infused) and (3) following the investigational agent infusion after successful PCI and stenting. There was no evidence of clinically important coronary microvascular obstruction related to infusion of the investigational agent.

If, for any reason, the site investigator withdrew a randomized participant prior to infusion of the investigational agent, the reason for early termination and data from the screening visit were entered into the eCRF by the study site. The participant did not remain in the study. If for any reason, a participant's study infusion was halted due to safety considerations, the participant remained in the study. A participant who prematurely withdrew from the study remained in the study for long-term safety follow-up.

Evaluation for safety was performed for up to 24 months post infusion for all non-Swedish sites. Participants enrolled in Sweden who consented for additional follow-up underwent safety assessments at 36, 48, and 60 months post-infusion of investigational agent. All participants were to have cardiac imaging using cardiac magnetic resonance imaging [cMRI] and 2D-echocardiography, Holter monitoring, clinical evaluations, and laboratory testing as outlined in the study protocol.

An independent Data Monitoring Safety Board (DSMB) reviewed all relevant acute peri-procedural data, serious adverse events (SAE), other adverse events (AE), and efficacy data (if requested) periodically until participant enrolment was closed.

ELIGIBILITY:
Key Inclusion Criteria:

* Clinical symptoms consistent with acute myocardial infarct (AMI) (pain, etc.) for a maximum of 12 hours from onset of symptoms to percutaneous coronary intervention (PCI).
* De Novo anterior AMI.
* Successful revascularization of the culprit lesion.

Key Exclusion Criteria:

* Prior AMI, known cardiomyopathy, or hospital admission for heart failure (HF).
* Significant valvular disease.
* Need for other interventional or surgical procedure to treat heart disease (planned or scheduled).
* Cardiogenic shock or hemodynamic instability within 24 hours of randomization.
* Prior PCI to LAD.
* Pacemaker, ICD (Implantable Cardioverter Defibrillator), or any other contra-indication for cardiac MRI.
* Prior or current participation in any stem cell study or any other investigational trial in the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2013-03-11 (Actual); Primary Completion 2021-04-06 (Actual); Study Completion 2021-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fred Grossman, DO, Study Director — Mesoblast, Inc.

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received matching-placebo solution 2 milliliter per minute (mL/min) infused Intracoronary for 60 min including line flush [0 Mesenchymal Precursor Cells (MPCs)/min] on Day 0.
Period: Overall Study
Arm/Group | Placebo | Mesenchymal Precursor Cells (MPC) 12.5 M | Mesenchymal Precursor Cells (MPC) 25 M
Started | 35 | 35 | 36
Completed | 32 | 28 | 32
Not Completed | 3 | 7 | 4
Not completed — Withdrawal of Consent | 0 | 3 | 1
Not completed — Lost to Follow-up | 1 | 1 | 1
Not completed — Adverse Event | 1 | 2 | 1
Not completed — Participants who were Randomized and Not Treated | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis population included all participants who were randomized, underwent percutaneous coronary intervention (PCI) and had infusion of study agent (mesenchymal precursor cells [MPCs] or placebo) initiated.
Groups:
- Placebo: Participants received matching-placebo solution 2 mL/min infused Intracoronary for 60 min including line flush [0 Mesenchymal Precursor Cells (MPCs)/min] on Day 0.
- Total: Total of all reporting groups
Arm/Group | Placebo | Mesenchymal Precursor Cells (MPC) 12.5 M | Mesenchymal Precursor Cells (MPC) 25 M | Total
Number analyzed (Participants) | 34 | 34 | 35 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (9.79) | 60.7 (13.11) | 57.6 (12.12) | 59.8 (11.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 8 | 17
  Male | 27 | 32 | 27 | 86
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 33 | 33 | 35 | 101
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 33 | 33 | 34 | 100
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 2
Left Ventricular (LV) End-systolic Volume (LVESV) as Assessed by Cardiac MRI [Mean (Standard Deviation); unit: milliliter (ml)] — Population: Full analysis population included all participants who were randomized, underwent PCI and had infusion of study product initiated as randomized. Number analyzed are the number of participants with data available for LVESV at Baseline. Baseline is defined as value measured at Day 2 to 4.
  milliliter (ml)
    number analyzed (Participants) | 30 | 28 | 32 | 90
    (all) | 85.544 (34.8935) | 91.728 (30.4476) | 92.163 (33.1251) | 89.821 (32.7025)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: Safety measure: An AE is any unfavorable and unintended sign, symptom, or disease, whether or not related to the investigational product. A TEAE was defined as any AE with onset post study drug treatment. An SAE was defined as any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is medically important.
Time Frame: Up to approximately 8 years
Population: The safety set included all participants who were randomly assigned to a treatment at screening and received treatment. Overall number analyzed is the participants available for analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Mesenchymal Precursor Cells (MPC) 12.5 M | Mesenchymal Precursor Cells (MPC) 25 M
Number analyzed (Participants) | 34 | 34 | 35
Participants
  TEAEs | 28 | 30 | 31
  SAEs | 14 | 16 | 14

ADVERSE EVENTS:
Time Frame: Up to approximately 8 years
Description: The safety set included all participants who were randomly assigned to a treatment at screening and received treatment.
Groups:
- Placebo: Participants received matching-placebo solution 2 mL/min infused Intracoronary for 60 mins including line flush [0 Mesenchymal Precursor Cells (MPCs)/min] on Day 0.
- Mesenchymal Precursor Cells (MPC) 12.5 M: Participants received MPC 12.5 solution 2 mL/min infused Intracoronary for 60 mins including line flush (2.5x10^5 MPCs/min) on Day 0.
- Mesenchymal Precursor Cells (MPC) 25 M: Participants received MPC 12.5 solution 2 mL/min infused Intracoronary for 60 mins including line flush (5.0x10^5 MPCs/min) on Day 0.
Arm/Group | Placebo | Mesenchymal Precursor Cells (MPC) 12.5 M | Mesenchymal Precursor Cells (MPC) 25 M
All-Cause Mortality (participants affected / at risk) | 0/34 | 2/34 | 2/35
Serious Adverse Events (participants affected / at risk) | 14/34 | 16/34 | 14/35
Other Adverse Events (participants affected / at risk) | 26/34 | 33/34 | 31/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=34) | Mesenchymal Precursor Cells (MPC) 12.5 M (N=34) | Mesenchymal Precursor Cells (MPC) 25 M (N=35)
Cardiac failure (Cardiac disorders) | 2 | 3 | 1
Angina pectoris (Cardiac disorders) | 2 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 1
Angina unstable (Cardiac disorders) | 1 | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 2 | 0 | 0
Cardiac ventricular thrombosis (Cardiac disorders) | 0 | 2 | 0
Coronary artery disease (Cardiac disorders) | 1 | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Arteriospasm coronary (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 1 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 1 | 3
Chest pain (General disorders) | 1 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 1 | 0
Vascular stent thrombosis (General disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 2 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 1
Diaphragmatic hernia gangrenous (Infections and infestations) | 1 | 0 | 0
Intervertebral discitis (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0
Migraine with aura (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 1 | 0
Acute psychosis (Psychiatric disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=34) | Mesenchymal Precursor Cells (MPC) 12.5 M (N=34) | Mesenchymal Precursor Cells (MPC) 25 M (N=35)
Ventricular tachycardia (Cardiac disorders) | 1 | 3 | 6
Bradycardia (Cardiac disorders) | 1 | 2 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 2 | 2
Palpitations (Cardiac disorders) | 0 | 3 | 1
Pericarditis (Cardiac disorders) | 0 | 1 | 3
Arteriospasm coronary (Cardiac disorders) | 2 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 2
Pyrexia (General disorders) | 5 | 2 | 3
Chest pain (General disorders) | 2 | 1 | 4
Fatigue (General disorders) | 2 | 3 | 1
Catheter site haematoma (General disorders) | 1 | 2 | 1
Oedema peripheral (General disorders) | 0 | 2 | 2
Multiple organ dysfunction syndrome (General disorders) | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 3 | 5
Nausea (Gastrointestinal disorders) | 1 | 5 | 3
Constipation (Gastrointestinal disorders) | 1 | 5 | 1
Vomiting (Gastrointestinal disorders) | 2 | 2 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 2 | 3
Influenza (Infections and infestations) | 2 | 1 | 1
Nasopharyngitis (Infections and infestations) | 3 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1 | 3
Urinary tract infection (Infections and infestations) | 1 | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 8 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Dizziness (Nervous system disorders) | 4 | 8 | 5
Headache (Nervous system disorders) | 2 | 1 | 2
Lethargy (Nervous system disorders) | 1 | 3 | 1
Dizziness postural (Nervous system disorders) | 1 | 2 | 0
Presyncope (Nervous system disorders) | 1 | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Hypotension (Vascular disorders) | 2 | 4 | 1
Hypertension (Vascular disorders) | 1 | 2 | 3
Peripheral coldness (Vascular disorders) | 1 | 4 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 3
Lower urinary tract symptoms (Renal and urinary disorders) | 0 | 2 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 4 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Blood triglycerides increased (Investigations) | 0 | 0 | 2
Anxiety (Psychiatric disorders) | 1 | 3 | 1
Insomnia (Psychiatric disorders) | 1 | 1 | 2
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0
Vision blurred (Eye disorders) | 0 | 2 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 2 | 0 | 2
Cardiac failure (Cardiac disorders) | 1 | 1 | 3
Angina pectoris (Cardiac disorders) | 2 | 3 | 1
Cardiac ventricular thrombosis (Cardiac disorders) | 1 | 4 | 0
Non-cardiac chest pain (General disorders) | 2 | 5 | 2
Pneumonia (Infections and infestations) | 0 | 2 | 1
Rales (Renal and urinary disorders) | 2 | 1 | 0
Dysphonia (Renal and urinary disorders) | 2 | 0 | 0

LIMITATIONS AND CAVEATS:
Originally, 225 de novo anterior STEMI participants were to undergo primary PCI. However, due to difficulty in consenting participants and operationalizing protocol under emergency conditions associated with acute STEMI, a major protocol amendment was required. The protocol was adjusted to randomize 105 participants. This 53% reduction in participants from the original protocol allowed preliminary evaluations of safety and feasibility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publications (abstracts, posters or presentations) must be presented to Publication Steering Committee for review prior to submission or public display and are not allowed prior to the publication of the primary manuscript, or eighteen (18) months from the conclusion of the Study. PI shall provide Sponsor a copy of any proposed public disclosure at least 30 days prior to submission. Sponsor may ask PI to delay the disclosure for a maximum of 60 days to file proprietary protection.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-04): https://cdn.clinicaltrials.gov/large-docs/90/NCT01781390/Prot_SAP_000.pdf